CLINICAL TRIAL: NCT02959944
Title: A Randomized, Double-Blind Phase 3 Study of Ibrutinib in Combination With Corticosteroids Versus Placebo in Combination With Corticosteroids in Subjects With New Onset Chronic Graft Versus Host Disease (cGVHD)
Brief Title: Ibrutinib in Combination With Corticosteroids vs Placebo in Combination With Corticosteroids in Participants With New Onset Chronic Graft Versus Host Disease (cGVHD)
Acronym: iNTEGRATE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PCYC-1140-IM
Record Dates: First submitted 2016-10-25; First posted 2016-11-09 (Estimated); Results first posted 2021-05-04 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Chronic Graft Versus Host Disease
Keywords: chronic graft versus host disease; PCYC1140; PCYC1140IM; 1140; Ibrutinib; GVHD; Steroid dependent; refractory; chronic; PCI32765; IMBRUVICA; Pharmacyclics; PCYC; graft versus host disease; immunology; new onset graft versus host disease; INTEGRATE; Corticosteroids; prednisone
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Graft vs Host Disease | interventions — ibrutinib; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ibrutinib + Prednisone (Experimental): Ibrutinib (420 mg) given orally once daily continuously starting on Week 1 Day 1 until cGVHD progression, progression of underlying malignancy, participant begins another systemic treatment for cGVHD or unacceptable toxicity. The 420 mg dose was adjusted for cytochrome P450 [CYP] inhibitors or hepatic dysfunction as applicable.
  Prednisone 1 mg/kg/d given orally once daily continuously starting on Week 1 Day 1 until unacceptable toxicity or until participant is successfully tapered from the prednisone. Starting prednisone dose may be as low as 0.5 mg/kg/d if a participant cannot tolerate higher doses.
  Interventions: Drug: ibrutinib; Drug: Prednisone
- Placebo + Prednisone (Placebo Comparator): Placebo given orally once daily continuously starting on Week 1 Day 1 until cGVHD progression, progression of underlying malignancy, participant begins another systemic treatment for cGVHD or unacceptable toxicity.
  Prednisone 1 mg/kg/d given orally once daily continuously starting on Week 1 Day 1 until unacceptable toxicity or until participant is successfully tapered from the prednisone. Starting prednisone dose may be as low as 0.5 mg/kg/d if a participant cannot tolerate higher doses.
  Interventions: Drug: Placebo; Drug: Prednisone

INTERVENTIONS:
Drug: ibrutinib — Ibrutinib capsules administered orally daily
  Other Names: IMBRUVICA®; PCI-32765
  Arms: Ibrutinib + Prednisone
Drug: Placebo — Placebo capsules administered orally daily
  Arms: Placebo + Prednisone
Drug: Prednisone — Prednisone administered daily

SUMMARY:
To evaluate the safety and efficacy of ibrutinib in combination with prednisone in subjects with newly diagnosed moderate to severe cGVHD.

ELIGIBILITY:
Key Inclusion Criteria:

* New onset moderate or severe cGVHD as defined by the 2014 National Institutes of Health (NIH) Consensus Development Project Criteria
* Need for systemic treatment with corticosteroids for cGVHD
* No previous systemic treatment for cGVHD (including extracorporeal photopheresis [ECP])
* Participants may be receiving other immunosuppressants for the prophylaxis or treatment of acute GVHD but if the subject is receiving prednisone for prophylaxis or treatment of acute GVHD it must be at or below 0.5 mg/kg/d
* Age ≥12 years old
* Karnofsky or Lansky (subjects <16 years) performance status ≥60

Key Exclusion Criteria:

* Received any previous systemic treatment for cGVHD with the exception of corticosteroids administered for cGVHD within the 72 hours prior to signing the informed consent form.
* Inability to begin a prednisone dose ≥0.5 mg/kg/d for the treatment of cGVHD
* Any uncontrolled infection or active infection requiring ongoing systemic treatment
* Progressive underlying malignant disease or any post-transplant lymphoproliferative disease
* Known bleeding disorders
* Active hepatitis C virus (HCV) or hepatitis B virus (HBV)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2020-03-27 (Actual); Study Completion 2021-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Justin Wahlstrom, MD, Study Director — Pharmacyclics LLC.
Locations (102):
- United States (38):
  - Arizona Oncology - Scottsdale - Cancer Transplant Institute Location /ID# 1140-1120, Scottsdale, Arizona
  - LPCH Stanford /ID# 1140-1128, Palo Alto, California
  - Ucsf /Id# 1140-0003, San Francisco, California
  - Stanford University/Stanford Cancer Center, Pasteur Drive /ID# 1140-0400, Stanford, California
  - UCHSC Anschultz Cancer Pavilion /ID# 1140-0068, Aurora, Colorado
  - Children's National Medical Center /ID# 1140-1122, Washington D.C., District of Columbia
  - Jackson Memorial Hospital, University of Miami /ID# 1140-0647, Miami, Florida
  - Florida Hospital Cancer Institute/Adventist Health System/Sunbelt, Inc /ID# 1140-1121, Orlando, Florida
  - Emory University, Winship Cancer Institute /ID# 1140-0033, Atlanta, Georgia
  - Emory University/Winship Cancer Institute /ID# 1140-1179, Atlanta, Georgia
  - University of Chicago /ID# 1140-0126, Chicago, Illinois
  - Loyola University /ID# 1140-0713, Maywood, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center /ID# 1140-0010, Indianapolis, Indiana
  - University of Kentucky /ID# 1140-1140, Lexington, Kentucky
  - University of Louisville Hospital /ID# 1140-1131, Louisville, Kentucky
  - University of Maryland /ID# 1140-0205, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center /ID# 1140-0020, Boston, Massachusetts
  - Boston Childrens Hospital /ID# 1140-1615, Boston, Massachusetts
  - Dana-Farber Cancer Institute /ID# 1140-0349, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer In /ID# 1140-0130, Detroit, Michigan
  - University of Minnesota /ID# 1140-0807, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, MN /ID# 1140-0240, Rochester, Minnesota
  - Hackensack University Medical Center/ John Theurer Cancer Center /ID# 1140-0343, Hackensack, New Jersey
  - Rutgers Cancer Institute of NJ /ID# 1140-0803, New Brunswick, New Jersey
  - New York Presbyterian Hospital/Weill Cornell Med College /ID# 1140-0200, New York, New York
  - Stony Brook University Medical Center /ID# 1140-0719, New York, New York
  - Columbia University Medical Center, MS-CHONY /ID# 1140-1124, New York, New York
  - Weill Cornell Physicians - Hematologic Malignancies & Bone Marrow Transplant /ID# 1140-0019, New York, New York
  - University of Rochester Cancer Center /ID# 1140-0127, Rochester, New York
  - Montefiore Medical Center - Moses Campus /ID# 1140-0120, The Bronx, New York
  - University of North Carolina - Lineberger Comprehensive Cancer Center /ID# 1140-1133, Chapel Hill, North Carolina
  - Univ Hosp Cleveland /ID# 1140-0941, Cleveland, Ohio
  - University of Pittsburgh - UPMC (Hillman Cancer Center) /ID# 1140-0050, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, MUSC /ID# 1140-0738, Charleston, South Carolina
  - Vanderbilt University Medical Center Vanderbilt Ingram Cancer Center /ID# 1140-0024, Nashville, Tennessee
  - Methodist San Antonio /ID# 1140-1118, San Antonio, Texas
  - Fred Hutchinson Cancer Research Center /ID# 1140-0404, Seattle, Washington
  - West Virginia University /ID# 1140-1090, Morgantown, West Virginia
- Australia (6):
  - The Kinghorn Cancer Centre /ID# 1140-1165, Darlinghurst, New South Wales
  - Westmead Hospital /ID# 1140-0848, Westmead, New South Wales
  - Royal Brisbane and Women's Hospital /ID# 1140-0190, Herston, Queensland
  - Royal Children's Hospital/ID# 1140-1154, Parkville, Victoria
  - Royal Melbourne Hospital (RMH) /ID# 1140-0633, Parkville, Victoria
  - Fiona Stanley Hospital /ID# 1140-0880, Perth, Western Australia
- Austria (2):
  - Univ. Klinik for Innere Medizin, Klinische Abteilung for Hematologie, Graz /ID# 1140-0373, Graz
  - Krankenhaus der Elisabethinen Linz /ID# 1140-0849, Linz
- Canada (4):
  - University of British Columbia (UBC) - Vancouver General Hospital (VGH) /ID# 1140-1166, Vancouver, British Columbia
  - The Ottawa Hospital Regional Cancer Center /ID# 1140-0159, Ottawa, Ontario
  - Princess Margaret Cancer Centre /ID# 1140-0043, Toronto, Ontario
  - CHU Sainte-Justine /ID# 1140-1143, Montreal, Quebec
- China (3):
  - The First Affiliated Hospital of Soochow University /ID# 1140-1208, Suzhou, Jiangsu
  - Chinese PLA General Hospital /ID# 1140-1198, Beijing
  - Nanfang Hospital /ID# 1140-1379, Guangzhou
- UHC Zagreb /ID# 1140-1169, Zagreb, Croatia
- France (7):
  - Hopital de Brabois /ID# 1140-0775, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - CHU Amiens Groupe hospitalier Sud /ID# 1140-1205, Amiens
  - CHU de GRENOBLE Alpes /ID# 1140-1058, Grenoble
  - Centre Hospitalier Regional Universitaire de Lille /ID# 1140-0750, Lille
  - CHU de Nantes /ID# 1140-0520, Nantes
  - Groupe Hospitalier Pitie-Salpetriere /ID# 1140-0918, Paris
  - Hopital Saint-Louis - Institut Hematologie Centre Hayem CHU /ID# 1140-0735, Paris, Île-de-France Region
- Germany (6):
  - Robert Bosch Hospital /ID# 1140-1160, Stuttgart, Baden-Wurttemberg
  - Universitatsklinikum Munster /ID# 1140-1195, Munster, Lower Saxony
  - Universitaetsklinikum Dresden /ID# 1140-1367, Dresden
  - Hannover Medical School /ID# 1140-1141, Hanover
  - Dr. Haunerschen Kinderspital /ID# 1140-1142, Munich
  - University Hospital of Regensburg /ID# 1140-1446, Regensburg
- St. Laszlo Hospital /ID# 1140-1164, Budapest, Hungary
- Italy (6):
  - IRCCS Ospedale Pediatrico Bambino Gesu /ID# 1140-1150, Rome, Lazio
  - A.O. Univ. Ospedali Riuniti /ID# 1140-0932, Ancona, The Marches
  - ASST Papa Giovanni XXIII /ID# 1140-1231, Bergamo
  - Ospedale San Raffaele IRCCS /ID# 1140-0523, Milan
  - University of Torino /ID# 1140-1268, Torino
  - Centro Trapianti Cellule Staminali, Ospedale Infantile Regina Margherita /ID# 1140-1156, Turin
- Japan (14):
  - Anjou Kousei Hospital /ID# 1140-1435, Anjo, Aichi-ken
  - Hiroshima Red Cross Hospital and Atomic-bomb Survivors Hospital /ID# 1140-1437, Hiroshima, Hiroshima
  - Kobe City Medical Center General Hospital /ID# 1140-1438, Kobe, Hyōgo
  - Hyogo College of Medicine College Hospital /Id# 1140-1434, Nishinomiya-shi, Hyōgo
  - Duplicate_University of Tsukuba Hospital /ID# 1140-1445, Tsukuba, Ibaraki
  - Tokai University Hospital /ID# 1140-1444, Isehara-shi, Kanagawa
  - Duplicate_Kurashiki Central Hospital /ID# 1140-1442, Kurishiki-shi, Okayama-ken
  - Okayama University Hospital /ID# 1140-1430, Okayama, Okayama-ken
  - Osaka Women's and Children's Hospital /ID# 1140-1440, Izumi-Shi, Osaka
  - Osaka City University Hospital /ID# 1140-1157, Osaka, Osaka
  - Dup_Tokyo Metropolitan Cancer and Infectious Diseases Center Komagome Hospital /ID# 1140-1439, Bunkyo-ku, Tokyo
  - National Center for Child Health and Development /ID# 1140-1443, Setagaya-ku, Tokyo
  - Kumamoto Medical Center /ID# 1140-1431, Kumamoto
  - Hokkaido University Hospital /ID# 1140-1436, Sapporo
- Singapore (2):
  - National University Cancer Institute - National University Health System /ID# 1140-1155, Singapore
  - Singapore General Hospital /ID# 1140-1162, Singapore
- South Korea (6):
  - Kyungpook National Univ Hosp /ID# 1140-1153, Daegu, Daegu Gwang Yeogsi
  - Yonsei University Health System, Severance Hospital /ID# 1140-0927, Seodaemun-gu, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 1140-0925, Seoul, Seoul Teugbyeolsi
  - Cath Univ Seoul St Mary's Hosp /ID# 1140-0928, Seoul, Seoul Teugbyeolsi
  - SoonChunHyang University Seoul /ID# 1140-1163, Seoul
  - Asan Medical Center /ID# 1140-0963, Seoul
- Spain (4):
  - Hospital Clinic /ID# 1140-0533, Barcelona
  - Hospital Santa Creu i Sant Pau /ID# 1140-0535, Barcelona
  - Hospital Universitario Virgen del Rocio /ID# 1140-0863, Seville
  - Hospital Clinico Universitario de Valencia /ID# 1140-1145, Valencia
- Taiwan (2):
  - China Medical University Hosp /ID# 1140-1199, Taichung, Taichung
  - National Taiwan Univ Hosp /ID# 1140-1184, Taipei City, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Requests for access to individual participant data from clinical studies conducted by Pharmacyclics LLC, an AbbVie Company, can be submitted through Yale Open Data Access (YODA) Project site at the following link.
URL: http://yoda.yale.edu

REFERENCES:
- [Derived] Miklos DB, Abu Zaid M, Cooney JP, Albring JC, Flowers M, Skarbnik AP, Yakoub-Agha I, Ko BS, Bruno B, Waller EK, Yared J, Sohn SK, Bulabois CE, Teshima T, Jacobsohn D, Greinix H, Mokatrin A, Lee Y, Wahlstrom JT, Styles L, Socie G. Ibrutinib for First-Line Treatment of Chronic Graft-Versus-Host Disease: Results From the Randomized Phase III iNTEGRATE Study. J Clin Oncol. 2023 Apr 1;41(10):1876-1887. doi: 10.1200/JCO.22.00509. Epub 2023 Jan 6. PMID 36608310

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 66 sites overall: 24 sites in North America, and 42 sites in the rest of the world.
Period: Overall Study
Arm/Group | Ibrutinib + Prednisone | Placebo + Prednisone
Started | 95 | 98
Received at Least 1 Dose of Study Drug | 94 | 96
Completed | 95 | 98
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ibrutinib + Prednisone: Ibrutinib (420 mg) given orally once daily continuously starting on Week 1 Day 1 until cGVHD progression, progression of underlying malignancy, participant begins another systemic treatment for cGVHD or unacceptable toxicity. The 420 mg dose was adjusted for CYP inhibitors or hepatic dysfunction as applicable.
  Prednisone 1 mg/kg/d given orally once daily continuously starting on Week 1 Day 1 until unacceptable toxicity or until participant is successfully tapered from the prednisone. Starting prednisone dose may be as low as 0.5 mg/kg/d if a participant cannot tolerate higher doses.
- Total: Total of all reporting groups
Arm/Group | Ibrutinib + Prednisone | Placebo + Prednisone | Total
Number analyzed (Participants) | 95 | 98 | 193
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.0 (14.48) | 51.1 (14.99) | 50.6 (14.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 33 | 67
  Male | 61 | 65 | 126
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 7
  Not Hispanic or Latino | 78 | 78 | 156
  Unknown or Not Reported | 12 | 18 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 27 | 19 | 46
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 6 | 4 | 10
  White | 47 | 58 | 105
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 12 | 16 | 28

OUTCOME MEASURES:

1. Primary Outcome: Primary Analysis: Response Rate at 48 Weeks
Description: Response rate was defined as the percentage of participants who were responders. Responders were defined as participants who had a complete response (CR) or a partial response (PR) at 48 weeks without starting any subsequent therapy for cGVHD or having evidence of relapse of their underlying disease that was indication for transplant prior to response assessment at 48 weeks.
  Response was defined using the National Institutes of Health (NIH) Consensus Panel Chronic GVHD Activity Assessment (2014). Skin, mouth, liver, upper and lower gastrointestinal, esophagus, lung, eye, and joint/fascia are the organs or sites considered in evaluating overall response. CR is defined as resolution of all manifestations in each organ or site. PR is defined as improvement in at least 1 organ or site without progression in any other organ or site.
Time Frame: 48 weeks (Cumulatively up to 30 March 2020)
Population: Intent to Treat Population: all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Ibrutinib + Prednisone | Placebo + Prednisone
Number analyzed (Participants) | 95 | 98
percentage of participants | 41.1 | 36.7
Statistical Analysis 1: Comparison: Ibrutinib + Prednisone vs Placebo + Prednisone; Test type: Superiority; p = 0.5384, Chi-squared — P-value is computed using non-stratified Chi-Square test; Difference in Rates = 0.043, 95% CI 2-sided [-0.094 to 0.181] — Confidence interval is computed using normal approximation

2. Primary Outcome: Final Analysis: Response Rate at 48 Weeks
Description: as for outcome 1
Time Frame: 48 weeks (Cumulatively up to 12 July 2021)
Population: Intent to Treat Population: all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Ibrutinib + Prednisone | Placebo + Prednisone
Number analyzed (Participants) | 95 | 98
percentage of participants | 41.1 | 36.7
Statistical Analysis 1: Comparison: Ibrutinib + Prednisone vs Placebo + Prednisone; Test type: Superiority; p = 0.5384, Chi-squared — P-value is computed using non-stratified Chi-Square test; Difference in Rates = 0.043, 95% CI 2-sided [-0.094 to 0.181] — Confidence interval is computed using normal approximation

3. Secondary Outcome: Primary Analysis: Cumulative Incidence of Withdrawal of All Corticosteroids for Treatment of cGVHD
Description: The cumulative incidence of withdrawal of all corticosteroids (95% confidence interval [CI]) was calculated using SAS lifetest procedure adjusting for competing risks including death, cGVHD progression, relapse of underlying disease, and start of subsequent cGVHD therapy. Data presented are the estimated proportion of participants withdrawing all corticosteroids at given time point. The time to withdrawal of corticosteroids is computed from randomization date to the first date of withdrawal of all corticosteroids for treatment of cGVHD to 0 mg daily for at least 30 days.
Time Frame: Months 3, 6, 9, 12, 15, 18, 21, 24 (Cumulatively up to 30 March 2020)
Population: Intent to Treat Population: all randomized participants. Participants with withdrawal of all corticosteroids. No participants were on corticosteroids at 21 and 24 Months in the Ibrutinib + Prednisone Arm/Group.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Ibrutinib + Prednisone | Placebo + Prednisone
Number analyzed (Participants) | 40 | 36
proportion of participants
  3 Months | 0.042 [0.014 to 0.097] | 0.021 [0.004 to 0.066]
  6 Months | 0.229 [0.149 to 0.320] | 0.216 [0.140 to 0.304]
  9 Months | 0.318 [0.225 to 0.415] | 0.322 [0.231 to 0.417]
  12 Months | 0.392 [0.290 to 0.492] | 0.356 [0.260 to 0.453]
  15 Months | 0.419 [0.314 to 0.520] | 0.356 [0.260 to 0.453]
  18 Months | 0.419 [0.314 to 0.520] | 0.356 [0.260 to 0.453]
  21 Months: number analyzed (Participants) | 0 | 36
  21 Months |  | 0.425 [0.299 to 0.545]
  24 Months: number analyzed (Participants) | 0 | 36
  24 Months |  | 0.425 [0.299 to 0.545]
Statistical Analysis 1: Comparison: Ibrutinib + Prednisone vs Placebo + Prednisone; Test type: Superiority; p = 0.324, Chi-squared — Gray's chi-square test (p-value) was calculated using SAS lifetest procedure adjusting for competing risks including death, cGVHD progression, relapse of underlying disease, and start of subsequent cGVHD therapy

4. Secondary Outcome: Final Analysis: Cumulative Incidence of Withdrawal of All Corticosteroids for Treatment of cGVHD
Description: as for outcome 3
Time Frame: Months 3, 6, 9, 12, 15, 18, 21, 24 (Cumulatively up to 12 July 2021)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Ibrutinib + Prednisone | Placebo + Prednisone
Number analyzed (Participants) | 45 | 38
proportion of participants
  3 Months | 0.042 [0.014 to 0.097] | 0.021 [0.004 to 0.066]
  6 Months | 0.218 [0.140 to 0.308] | 0.219 [0.142 to 0.307]
  9 Months | 0.318 [0.225 to 0.414] | 0.326 [0.234 to 0.422]
  12 Months | 0.406 [0.305 to 0.505] | 0.359 [0.263 to 0.455]
  15 Months | 0.439 [0.336 to 0.538] | 0.359 [0.263 to 0.455]
  18 Months | 0.450 [0.346 to 0.549] | 0.369 [0.272 to 0.466]
  21 Months | 0.495 [0.388 to 0.593] | 0.391 [0.292 to 0.489]
  24 Months | 0.495 [0.388 to 0.593] | 0.391 [0.292 to 0.489]
Statistical Analysis 1: Comparison: Ibrutinib + Prednisone vs Placebo + Prednisone; Test type: Superiority; p = 0.281, Chi-squared — [p-value comment as in outcome 3, analysis 1]

5. Secondary Outcome: Primary Analysis: Cumulative Incidence of Withdrawal of All Immunosuppressants
Description: The cumulative incidence of withdrawal of all immunosuppressants (95% CI) was calculated using SAS lifetest procedure adjusting for competing risks including death, cGVHD progression, relapse of underlying disease, and start of subsequent cGVHD therapy. Data presented are the estimated proportion of participants withdrawing all immunosuppressants at a given time point. The time to withdrawal of all immunosuppressants is computed from randomization date to the first date of withdrawal of all immunosuppressants for treatment of cGVHD, sustained for at least 30 days. All immunosuppressants include corticosteroids but they do not include ibrutinib.
Time Frame: Months 3, 6, 9, 12, 15, 18, 21, 24 (cumulatively up to 30 March 2020)
Population: Intent to Treat Population: all randomized participants. Participants with withdrawal of all immunosuppressants
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Ibrutinib + Prednisone | Placebo + Prednisone
Number analyzed (Participants) | 29 | 24
proportion of participants
  3 Months | 0.011 [0.001 to 0.052] | 0.000 [NA to NA] — At the time of primary analysis, the 95% confidence interval for the median could not be estimated because the data was skewed.
  6 Months | 0.142 [0.079 to 0.222] | 0.134 [0.075 to 0.210]
  9 Months | 0.220 [0.141 to 0.310] | 0.207 [0.132 to 0.294]
  12 Months | 0.256 [0.170 to 0.350] | 0.241 [0.160 to 0.331]
  15 Months | 0.285 [0.193 to 0.383] | 0.241 [0.160 to 0.331]
  18 Months | 0.313 [0.210 to 0.422] | 0.241 [0.160 to 0.331]
  21 Months | 0.376 [0.252 to 0.499] | 0.268 [0.174 to 0.370]
  24 Months | 0.421 [0.280 to 0.556] | 0.268 [0.174 to 0.370]
Statistical Analysis 1: Comparison: Ibrutinib + Prednisone vs Placebo + Prednisone; Test type: Superiority; p = 0.275, Chi-squared — [p-value comment as in outcome 3, analysis 1]

6. Secondary Outcome: Final Analysis: Cumulative Incidence of Withdrawal of All Immunosuppressants
Description: as for outcome 5
Time Frame: Months 3, 6, 9, 12, 15, 18, 21, 24 (Cumulatively up to 12 July 2021)
Population: Intent to Treat Population: all randomized participants. Participants with withdrawal of all immunosuppressants
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Ibrutinib + Prednisone | Placebo + Prednisone
Number analyzed (Participants) | 37 | 30
proportion of participants
  3 Months | 0.011 [0.001 to 0.052] | 0.000 [NA to NA] — At the time of primary analysis, the 95% confidence interval for the median could not be estimated because the data was skewed.
  6 Months | 0.143 [0.080 to 0.224] | 0.136 [0.076 to 0.213]
  9 Months | 0.222 [0.142 to 0.313] | 0.221 [0.143 to 0.309]
  12 Months | 0.280 [0.191 to 0.375] | 0.264 [0.179 to 0.356]
  15 Months | 0.314 [0.220 to 0.412] | 0.274 [0.188 to 0.367]
  18 Months | 0.349 [0.251 to 0.448] | 0.285 [0.197 to 0.379]
  21 Months | 0.372 [0.272 to 0.472] | 0.307 [0.216 to 0.402]
  24 Months | 0.406 [0.303 to 0.507] | 0.307 [0.216 to 0.402]
Statistical Analysis 1: Comparison: Ibrutinib + Prednisone vs Placebo + Prednisone; Test type: Superiority; p = 0.216, Chi-squared — [p-value comment as in outcome 3, analysis 1]

7. Secondary Outcome: Primary Analysis: Response Rate at 24 Weeks
Description: Response rate was defined as the percentage of participants who were responders. Responders were defined as participants who had a CR or PR at 24 weeks without starting any subsequent therapy for cGVHD or having evidence of relapse of their underlying disease that was indication for transplant prior to response assessment at 24 weeks.
  Response was defined using the National Institutes of Health (NIH) Consensus Panel Chronic GVHD Activity Assessment (2014). Skin, mouth, liver, upper and lower gastrointestinal, esophagus, lung, eye, and joint/fascia are the organs or sites considered in evaluating overall response. CR is defined as resolution of all manifestations in each organ or site. PR is defined as improvement in at least 1 organ or site without progression in any other organ or site.
Time Frame: 24 weeks (Cumulatively up to 30 March 2020)
Population: Intent to Treat Population: all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Ibrutinib + Prednisone | Placebo + Prednisone
Number analyzed (Participants) | 95 | 98
percentage of participants | 47.4 | 54.1
Statistical Analysis 1: Comparison: Ibrutinib + Prednisone vs Placebo + Prednisone; Test type: Superiority; p = 0.3510, Chi-squared — P-value was computed using non-stratified Chi-Square test; Difference in Rates = -0.067, 95% CI 2-sided [-0.208 to 0.074] — Confidence interval is computed using normal approximation

8. Secondary Outcome: Final Analysis: Response Rate at 24 Weeks
Description: as for outcome 7
Time Frame: 24 weeks (Cumulatively up to 12 July 2021)
Population: Intent to Treat Population: all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Ibrutinib + Prednisone | Placebo + Prednisone
Number analyzed (Participants) | 95 | 98
percentage of participants | 47.4 | 54.1
Statistical Analysis 1: Comparison: Ibrutinib + Prednisone vs Placebo + Prednisone; Test type: Superiority; p = 0.3510, Chi-squared — P-value was computed using non-stratified Chi-Square test; Difference in Rates = -0.067, 95% CI 2-sided [-0.208 to 0.074] — Confidence interval is computed using normal approximation

9. Secondary Outcome: Primary Analysis: Percentage of Participants With Improvement in Overall Score on Lee cGVHD Symptom Scale at Two Consecutive Visits
Description: Clinically meaningful improvement on Lee cGVHD symptom scale was defined as at least a 7-point decrease in Lee Symptom Scale overall summary score on at least 2 consecutive visits, not preceded by progressive disease, relapse of underlying disease or start of subsequent cGVHD treatment.
  The Lee cGVHD Symptom Scale score has 7 subscales (Skin, Eyes and Mouth, Breathing, Eating and Digestion, Muscles and Joints, Energy, and Mental and Emotional) with ratings as follows: 0- Not at all, 1- Slightly, 2 Moderately, 3 Quite a bit, 4-Extremely, with lower values representing a better outcome. A score is calculated for each subscale by taking the mean of all items completed if more than 50% were answered and normalizing to a 0 to 100 scale. An overall score is calculated as the average of these 7 subscales if at least 4 subscales have valid scores.
Time Frame: Assessed at Weeks 5, 13, 25, 37, 49, 30 days after the last dose of study drug, and then every 12 weeks of follow-up until progressed disease. (Cumulatively up to 30 March 2020)
Population: Intent to Treat Population: all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Ibrutinib + Prednisone | Placebo + Prednisone
Number analyzed (Participants) | 95 | 98
percentage of participants | 38.9 | 26.5
Statistical Analysis 1: Comparison: Ibrutinib + Prednisone vs Placebo + Prednisone; Test type: Superiority; p = 0.0659, Chi-squared — P-value is computed using non-stratified Chi-Square test; Difference in Rates = 0.124, 95% CI 2-sided [-0.007 to 0.256] — Confidence interval is computed using normal approximation

10. Secondary Outcome: Final Analysis: Percentage of Participants With Improvement in Overall Score on Lee cGVHD Symptom Scale at Two Consecutive Visits
Description: as for outcome 9
Time Frame: Assessed at Weeks 5, 13, 25, 37, 49, 30 days after the last dose of study drug, and then every 12 weeks of follow-up until progressed disease. (Cumulatively up to 12 July 2021)
Population: Intent to Treat Population: all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Ibrutinib + Prednisone | Placebo + Prednisone
Number analyzed (Participants) | 95 | 98
percentage of participants | 43.2 | 30.6
Statistical Analysis 1: Comparison: Ibrutinib + Prednisone vs Placebo + Prednisone; Test type: Superiority; p = 0.0708, Chi-squared — P-value is computed using non-stratified Chi-Square test; Difference in Rates = 0.125, 95% CI 2-sided [-0.010 to 0.261]

11. Secondary Outcome: Primary Analysis: Percentage of Participants Who Achieved Reduction of Prednisone Dose Level to Less Than 0.15 mg/kg/Day at 24 Weeks Sustained for at Least 30 Days
Time Frame: 24 weeks (Cumulatively up to 30 March 2020)
Population: Intent to Treat Population: all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Ibrutinib + Prednisone | Placebo + Prednisone
Number analyzed (Participants) | 95 | 98
percentage of participants | 40.0 | 45.9
Statistical Analysis 1: Comparison: Ibrutinib + Prednisone vs Placebo + Prednisone; Test type: Superiority; p = 0.4064, Chi-squared — P-value was computed using non-stratified Chi-Square test; Difference in Rates = -0.059, 95% CI 2-sided [-0.199 to 0.080] — Confidence interval was computed using normal approximation

12. Secondary Outcome: Final Analysis: Percentage of Participants Who Achieved Reduction of Prednisone Dose Level to Less Than 0.15 mg/kg/Day at 24 Weeks Sustained for at Least 30 Days
Time Frame: 24 weeks (Cumulatively up to 12 July 2021)
Population: Intent to Treat Population: all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Ibrutinib + Prednisone | Placebo + Prednisone
Number analyzed (Participants) | 95 | 98
percentage of participants | 41.1 | 45.9
Statistical Analysis 1: Comparison: Ibrutinib + Prednisone vs Placebo + Prednisone; Test type: Superiority; p = 0.4955, Chi-squared — P-value was computed using non-stratified Chi-Square test; Difference in Rates = -0.049, 95% CI 2-sided [-0.188 to 0.091] — Confidence interval was computed using normal approximation

13. Secondary Outcome: Primary Analysis: Overall Survival (OS)
Description: OS was defined as the time of randomization until the time of death due to any cause, in months.
Time Frame: Median time on study (cumulatively up to 30 March 2020) was 19.8 months and 18.4 months for the Ibrutinib + Prednisone and Placebo + Prednisone arms, respectively.
Population: Intent to Treat Population: all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ibrutinib + Prednisone | Placebo + Prednisone
Number analyzed (Participants) | 95 | 98
months | NA [30.0 to NA] — Not estimable due to the low number of events accrued by data cutoff. | NA [NA to NA] — Not estimable due to the low number of events accrued by data cutoff.
Statistical Analysis 1: Comparison: Ibrutinib + Prednisone vs Placebo + Prednisone; Test type: Superiority; Hazard Ratio (HR) = 0.994, 95% CI 2-sided [0.507 to 1.949] — Hazard ratio is estimated using unstratified Cox regression model with treatment as the only covariate

14. Secondary Outcome: Final Analysis: OS
Description: OS was defined as the time of randomization until the time of death due to any cause, in months.
Time Frame: Median time on study (cumulatively up to 12 July 2021) was 33.1 months and 32.5 months for the Ibrutinib + Prednisone and Placebo + Prednisone arms, respectively.
Population: Intent to Treat Population: all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ibrutinib + Prednisone | Placebo + Prednisone
Number analyzed (Participants) | 95 | 98
months | NA [NA to NA] — Not estimable due to the low number of events accrued by data cutoff. | NA [NA to NA] — Not estimable due to the low number of events accrued by data cutoff.
Statistical Analysis 1: Comparison: Ibrutinib + Prednisone vs Placebo + Prednisone; Test type: Superiority; Hazard Ratio (HR) = 1.061, 95% CI 2-sided [0.591 to 1.904] — Hazard ratio is estimated using unstratified Cox regression model with treatment as the only covariate

15. Secondary Outcome: Primary Analysis: Duration of Response (DOR) for Participants Who Had PR or CR at Any Time
Description: Response was defined using the NIH Consensus Panel Chronic GVHD Activity Assessment (2014). Skin, mouth, liver, upper and lower GI, esophagus, lung, eye, and joint/fascia are the organs or sites considered in evaluating overall response. CR was defined as resolution of all manifestations in each organ or site. PR was defined as improvement in at least 1 organ or site without progression in any other organ or site. Duration of response was estimated by Kaplan-Meier methodology.
Time Frame: Response was assessed every 4 weeks from Week 5 through Week 25, Week 37, Week 49, 30 days after the last dose of study drug, and then every 12 weeks of follow-up until progressed disease. (Cumulatively up to 30 March 2020)
Population: Participants in the Intent-to-Treat Population (all randomized participants) who had response of CR/PR at any time during the study and had not started any subsequent therapy for cGVHD or had evidence of relapse of their underlying disease that was indication for transplant at the time of response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ibrutinib + Prednisone | Placebo + Prednisone
Number analyzed (Participants) | 74 | 80
months | 19.8 [7.4 to NA] — At the time of primary analysis, the upper bound of 95% confidence interval for the median could not be estimated because the data was skewed. | 10.0 [6.5 to 13.1]
Statistical Analysis 1: Comparison: Ibrutinib + Prednisone vs Placebo + Prednisone; Test type: Superiority; p = 0.1010, Regression, Cox; Hazard Ratio (HR) = 0.697, 95% CI 2-sided [0.451 to 1.076]

16. Secondary Outcome: Final Analysis: DOR for Participants Who Had PR or CR at Any Time
Description: as for outcome 15
Time Frame: Response was assessed every 4 weeks from Week 5 through Week 25, Week 37, Week 49, 30 days after the last dose of study drug, and then every 12 weeks of follow-up until progressed disease. (Cumulatively up to 12 July 2021)
Population: as for outcome 15
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ibrutinib + Prednisone | Placebo + Prednisone
Number analyzed (Participants) | 74 | 80
months | 19.1 [7.4 to NA] — At the time of final analysis, the upper bound of 95% confidence interval for the median could not be estimated because the data was skewed. | 10.2 [6.5 to 17.1]
Statistical Analysis 1: Comparison: Ibrutinib + Prednisone vs Placebo + Prednisone; Test type: Superiority; p = 0.1004, Regression, Cox; Hazard Ratio (HR) = 0.717, 95% CI 2-sided [0.482 to 1.068]

17. Secondary Outcome: Primary Analysis: Number of Participants With Treatment-Emergent Adverse Events (AEs), Serious AEs (SAEs), and Discontinuations Due to AEs Placebo in Combination With Prednisone
Description: AE: any untoward medical occurrence, which does not necessarily have a causal relationship with this treatment. SAE: any untoward medical occurrence that at any dose: results in death; is life-threatening; requires in-patient hospitalization >24 hours or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is an important medical event. Severity was graded according to the Common Terminology Criteria for Adverse Events version 4.03 (grade 1=mild, grade 2=moderate, grade 3=severe, grade 4=life-threatening, grade 5=death). Treatment-related events are those that were possibly related or related to study treatment per investigator's judgment. Treatment emergent AEs (TEAEs) occurred from the first dose of study drug up to 30 days after the last dose of study drug.
Time Frame: From first dose of study drug through the end of treatment plus 30 days. As of data cutoff (cumulatively up to 30 March 2020), median ibrutinib treatment duration was 5.4 months and the median placebo treatment duration was 6.4 months.
Population: Safety Population: all participants who received at least one dose of either ibrutinib or placebo, analyzed according to the actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrutinib + Prednisone | Placebo + Prednisone
Number analyzed (Participants) | 94 | 96
Participants
  Any TEAE | 93 | 95
  Any Grade ≥ 3 TEAE | 60 | 64
  Any Ibrutinib-/Placebo-Related TEAE | 66 | 58
  Any Grade ≥ 3 Ibrutinib-/Placebo-Related TEAE | 32 | 28
  Any Corticosteroid-Related TEAE | 71 | 77
  Any Grade ≥ 3 Corticosteroid-Related TEAE | 32 | 36
  Any TEAE Leading to Discontinuation (DC) of Any Treatment | 21 | 24
  Any TEAE Leading to DC of Ibrutinib/Placebo | 21 | 23
  Any TEAE Leading to DC of Corticosteroid | 8 | 8
  Any Treatment Emergent SAE (TESAE) | 46 | 48
  Any Grade ≥ 3 TESAE | 43 | 46
  Any Treatment-Related TESAE | 27 | 28
  Any Ibrutinib/Placebo Treatment-Related TESAE | 24 | 19
  Any Corticosteroid Treatment-Related TESAE | 24 | 27
  Any Fatal TEAE | 10 | 7

18. Secondary Outcome: Final Analysis: Number of Participants With Treatment-Emergent Adverse Events (AEs), Serious AEs (SAEs), and Discontinuations Due to AEs Placebo in Combination With Prednisone
Description: as for outcome 17
Time Frame: From first dose of study drug through the end of treatment plus 30 days. As of data cutoff (cumulatively up to 12 July 2021), median ibrutinib treatment duration was 5.4 months and the median placebo treatment duration was 6.4 months.
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrutinib + Prednisone | Placebo + Prednisone
Number analyzed (Participants) | 94 | 96
Participants
  Any TEAE | 93 | 95
  Any Grade ≥ 3 TEAE | 64 | 64
  Any Ibrutinib-/Placebo-Related TEAE | 67 | 57
  Any Grade ≥ 3 Ibrutinib-/Placebo-Related TEAE | 35 | 27
  Any Corticosteroid-Related TEAE | 72 | 76
  Any Grade ≥ 3 Corticosteroid-Related TEAE | 34 | 35
  Any TEAE Leading to Discontinuation (DC) of Any Treatment | 23 | 28
  Any TEAE Leading to DC of Ibrutinib/Placebo | 22 | 27
  Any TEAE Leading to DC of Corticosteroid | 10 | 9
  Any Treatment Emergent SAE (TESAE) | 49 | 47
  Any Grade ≥ 3 TESAE | 46 | 45
  Any Treatment-Related TESAE | 29 | 27
  Any Ibrutinib/Placebo Treatment-Related TESAE | 26 | 18
  Any Corticosteroid Treatment-Related TESAE | 26 | 26
  Any Fatal TEAE | 12 | 6

ADVERSE EVENTS:
Time Frame: From first dose of study drug through the end of treatment plus 30 days. As of data cutoff (cumulatively up to 12 July 2021), median ibrutinib treatment duration was 5.4 months and the median placebo treatment duration was 6.4 months.
Groups:
- Ibrutinib: Ibrutinib (420 mg) given orally once daily continuously starting on Week 1 Day 1 until cGVHD progression, progression of underlying malignancy, participant begins another systemic treatment for cGVHD or unacceptable toxicity. The 420 mg dose was adjusted for cytochrome P450 [CYP] inhibitors or hepatic dysfunction as applicable.
  Prednisone 1 mg/kg/d given orally once daily continuously starting on Week 1 Day 1 until unacceptable toxicity or until participant is successfully tapered from the prednisone. Starting prednisone dose may be as low as 0.5 mg/kg/d if a participant cannot tolerate higher doses.
- Placebo: Placebo given orally once daily continuously starting on Week 1 Day 1 until cGVHD progression, progression of underlying malignancy, participant begins another systemic treatment for cGVHD or unacceptable toxicity.
  Prednisone 1 mg/kg/d given orally once daily continuously starting on Week 1 Day 1 until unacceptable toxicity or until participant is successfully tapered from the prednisone. Starting prednisone dose may be as low as 0.5 mg/kg/d if a participant cannot tolerate higher doses.
Arm/Group | Ibrutinib | Placebo
All-Cause Mortality (participants affected / at risk) | 23/94 | 22/96
Serious Adverse Events (participants affected / at risk) | 51/94 | 49/96
Other Adverse Events (participants affected / at risk) | 88/94 | 92/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibrutinib (N=94) | Placebo (N=96)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
COAGULOPATHY (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
THROMBOTIC MICROANGIOPATHY (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 (0) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 2 (2)
ATRIAL FLUTTER (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 1 (1) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 1 (1) | 1 (1)
MYOCARDITIS (Cardiac disorders) | 1 (1) | 0 (0)
PERICARDIAL EFFUSION (Cardiac disorders) | 2 (2) | 0 (0)
DIPLOPIA (Eye disorders) | 1 (1) | 0 (0)
COLITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 2 (2) | 1 (2)
ENTERITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 2 (2)
ILEUS (Gastrointestinal disorders) | 1 (1) | 0 (0)
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
MELAENA (Gastrointestinal disorders) | 1 (1) | 0 (0)
PANCREATIC ENZYME ABNORMALITY (Gastrointestinal disorders) | 1 (1) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1) | 0 (0)
DEATH (General disorders) | 2 (2) | 0 (0)
MALAISE (General disorders) | 1 (1) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 1 (1) | 3 (3)
CHOLECYSTITIS (Hepatobiliary disorders) | 1 (1) | 1 (1)
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
GRAFT VERSUS HOST DISEASE (Immune system disorders) | 0 (0) | 3 (3)
CHRONIC GRAFT VERSUS HOST DISEASE (Immune system disorders) | 3 (3) | 3 (3)
HYPOGAMMAGLOBULINAEMIA (Immune system disorders) | 1 (1) | 0 (0)
BACTERAEMIA (Infections and infestations) | 1 (1) | 1 (1)
BRONCHITIS (Infections and infestations) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0)
CELLULITIS (Infections and infestations) | 3 (3) | 0 (0)
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 0 (0) | 1 (2)
CYTOMEGALOVIRUS COLITIS (Infections and infestations) | 0 (0) | 1 (1)
CYTOMEGALOVIRUS INFECTION REACTIVATION (Infections and infestations) | 1 (1) | 1 (1)
DACRYOCYSTITIS (Infections and infestations) | 1 (1) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 1 (1) | 0 (0)
ENCEPHALITIS (Infections and infestations) | 1 (1) | 0 (0)
EPSTEIN-BARR VIRUS INFECTION REACTIVATION (Infections and infestations) | 1 (1) | 0 (0)
EYE INFECTION (Infections and infestations) | 0 (0) | 1 (1)
HAEMOPHILUS INFECTION (Infections and infestations) | 0 (0) | 1 (1)
INFLUENZA (Infections and infestations) | 4 (4) | 4 (4)
KLEBSIELLA BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0)
KLEBSIELLA SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
MASTOIDITIS (Infections and infestations) | 1 (1) | 0 (0)
MEDIASTINITIS (Infections and infestations) | 1 (1) | 0 (0)
METAPNEUMOVIRUS INFECTION (Infections and infestations) | 0 (0) | 1 (1)
PARAINFLUENZAE VIRUS INFECTION (Infections and infestations) | 1 (1) | 1 (1)
PAROTITIS (Infections and infestations) | 0 (0) | 1 (1)
PERIORBITAL CELLULITIS (Infections and infestations) | 1 (1) | 0 (0)
PERITONITIS (Infections and infestations) | 0 (0) | 1 (1)
PNEUMOCYSTIS JIROVECII PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 6 (8) | 9 (10)
PNEUMONIA CYTOMEGALOVIRAL (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA FUNGAL (Infections and infestations) | 1 (2) | 0 (0)
PNEUMONIA LEGIONELLA (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA PARAINFLUENZAE VIRAL (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA VIRAL (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA RESPIRATORY SYNCYTIAL VIRAL (Infections and infestations) | 0 (0) | 2 (2)
RESPIRATORY SYNCYTIAL VIRUS INFECTION (Infections and infestations) | 0 (0) | 1 (1)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 1 (1) | 2 (2)
SEPTIC SHOCK (Infections and infestations) | 2 (2) | 1 (1)
SINUSITIS (Infections and infestations) | 0 (0) | 1 (1)
SINUSITIS FUNGAL (Infections and infestations) | 1 (1) | 0 (0)
SKIN INFECTION (Infections and infestations) | 0 (0) | 1 (1)
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1)
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 1 (1)
URINARY TRACT INFECTION BACTERIAL (Infections and infestations) | 1 (1) | 0 (0)
UROSEPSIS (Infections and infestations) | 1 (1) | 0 (0)
WOUND INFECTION (Infections and infestations) | 1 (1) | 0 (0)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (1)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 1 (1) | 0 (0)
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
STEROID DIABETES (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
MUSCLE ATROPHY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MYOPATHY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
ACUTE MYELOID LEUKAEMIA RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4)
ACUTE PROMYELOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BENIGN NEOPLASM OF TESTIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
LEUKAEMIA RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
POST TRANSPLANT LYMPHOPROLIFERATIVE DISORDER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
PRIMARY MYELOFIBROSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
ISCHAEMIC STROKE (Nervous system disorders) | 1 (1) | 0 (0)
POSTERIOR REVERSIBLE ENCEPHALOPATHY SYNDROME (Nervous system disorders) | 1 (1) | 0 (0)
SEIZURE (Nervous system disorders) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 2 (2) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 1 (1)
MANIA (Psychiatric disorders) | 1 (1) | 0 (0)
SUBSTANCE-INDUCED PSYCHOTIC DISORDER (Psychiatric disorders) | 0 (0) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (2) | 2 (2)
CYSTITIS HAEMORRHAGIC (Renal and urinary disorders) | 0 (0) | 1 (1)
HAEMATURIA (Renal and urinary disorders) | 2 (2) | 0 (0)
HYDRONEPHROSIS (Renal and urinary disorders) | 1 (1) | 1 (1)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 1 (1)
OBSTRUCTIVE NEPHROPATHY (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 1 (1)
URETEROLITHIASIS (Renal and urinary disorders) | 1 (1) | 1 (1)
URETHRAL STENOSIS (Renal and urinary disorders) | 0 (0) | 1 (1)
INTERMENSTRUAL BLEEDING (Reproductive system and breast disorders) | 0 (0) | 1 (1)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
SCROTAL OEDEMA (Reproductive system and breast disorders) | 0 (0) | 1 (1)
BRONCHITIS CHRONIC (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY MASS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 2 (2)
PHLEBITIS (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibrutinib (N=94) | Placebo (N=96)
INCREASED TENDENCY TO BRUISE (Blood and lymphatic system disorders) | 9 (10) | 8 (8)
ANAEMIA (Blood and lymphatic system disorders) | 4 (17) | 11 (21)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 6 (11)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 18 (30) | 15 (25)
PALPITATIONS (Cardiac disorders) | 5 (5) | 3 (3)
CUSHINGOID (Endocrine disorders) | 3 (3) | 6 (6)
CATARACT (Eye disorders) | 2 (3) | 7 (8)
DRY EYE (Eye disorders) | 5 (6) | 4 (4)
VISION BLURRED (Eye disorders) | 7 (7) | 9 (10)
ABDOMINAL PAIN (Gastrointestinal disorders) | 8 (10) | 6 (6)
CONSTIPATION (Gastrointestinal disorders) | 7 (7) | 14 (15)
DIARRHOEA (Gastrointestinal disorders) | 14 (20) | 13 (19)
DYSPEPSIA (Gastrointestinal disorders) | 7 (7) | 4 (4)
NAUSEA (Gastrointestinal disorders) | 13 (20) | 13 (15)
VOMITING (Gastrointestinal disorders) | 15 (20) | 8 (8)
ASTHENIA (General disorders) | 5 (7) | 6 (7)
FATIGUE (General disorders) | 17 (22) | 18 (30)
INFLUENZA LIKE ILLNESS (General disorders) | 5 (6) | 1 (1)
OEDEMA PERIPHERAL (General disorders) | 25 (37) | 13 (17)
PYREXIA (General disorders) | 7 (7) | 16 (22)
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 6 (19) | 6 (10)
HYPOGAMMAGLOBULINAEMIA (Immune system disorders) | 5 (5) | 3 (3)
BRONCHITIS (Infections and infestations) | 2 (2) | 7 (8)
CONJUNCTIVITIS (Infections and infestations) | 4 (5) | 5 (6)
HERPES ZOSTER (Infections and infestations) | 5 (6) | 5 (5)
INFLUENZA (Infections and infestations) | 5 (5) | 6 (7)
NASOPHARYNGITIS (Infections and infestations) | 6 (6) | 8 (11)
PARONYCHIA (Infections and infestations) | 5 (5) | 2 (2)
RHINOVIRUS INFECTION (Infections and infestations) | 1 (1) | 7 (7)
SINUSITIS (Infections and infestations) | 1 (1) | 5 (8)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 15 (24) | 15 (21)
CONTUSION (Injury, poisoning and procedural complications) | 10 (11) | 4 (5)
FALL (Injury, poisoning and procedural complications) | 3 (4) | 7 (7)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 7 (11) | 16 (29)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 13 (17)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 3 (3) | 6 (12)
BLOOD CREATININE INCREASED (Investigations) | 5 (8) | 6 (7)
PLATELET COUNT DECREASED (Investigations) | 7 (13) | 6 (10)
WEIGHT DECREASED (Investigations) | 6 (6) | 4 (4)
WEIGHT INCREASED (Investigations) | 5 (7) | 6 (6)
DECREASED APPETITE (Metabolism and nutrition disorders) | 7 (8) | 7 (8)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 3 (3) | 8 (10)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 4 (6) | 13 (23)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 11 (21) | 14 (21)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 4 (10) | 8 (11)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 9 (10) | 6 (9)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 3 (5) | 9 (11)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 12 (19) | 13 (16)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 6 (7) | 11 (12)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 5 (7) | 9 (9)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 17 (20) | 16 (27)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (6)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 5 (6) | 5 (5)
DIZZINESS (Nervous system disorders) | 10 (10) | 11 (16)
HEADACHE (Nervous system disorders) | 13 (19) | 12 (17)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 6 (7) | 2 (5)
TREMOR (Nervous system disorders) | 5 (5) | 9 (10)
ANXIETY (Psychiatric disorders) | 5 (5) | 7 (8)
DEPRESSION (Psychiatric disorders) | 5 (6) | 2 (2)
INSOMNIA (Psychiatric disorders) | 26 (28) | 18 (20)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 3 (7) | 8 (9)
COUGH (Respiratory, thoracic and mediastinal disorders) | 21 (24) | 29 (37)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 9 (12) | 14 (16)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (6)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 4 (5)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 3 (3)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 5 (8) | 3 (3)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 8 (8)
PRURITUS (Skin and subcutaneous tissue disorders) | 6 (7) | 7 (10)
HYPERTENSION (Vascular disorders) | 10 (16) | 13 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
1. Institution/Investigator will not publish without Sponsor prior review and approval
2. Institution/Investigator will not publish until the earlier of (i) results of study are submitted for publication (ii) notification that submission of the multicenter results are no longer planned (iii) 18 months after study termination.

DOCUMENTS (2):
  • Study Protocol (2019-02-06): https://cdn.clinicaltrials.gov/large-docs/44/NCT02959944/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-28): https://cdn.clinicaltrials.gov/large-docs/44/NCT02959944/SAP_001.pdf